CLINICAL TRIAL: NCT00814424
Title: Quantitive And Qualitive Assessment Of The Oxygen Delivery And EtCO2 Sampling With The Smart Bite Block Mark III During An Upper Endoscopic Procedure Under Sedation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Oridion (Industry)
Responsible Party: David Gozal MD, Director of Sedation, Hadassah Medical Center, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0452-08-HMO
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2008-12-24 (Estimated); Status verified 2008-12

CONDITIONS: Ventilatory Status of Deeply Sedated ERCP Patients
Keywords: EtCO2; supplemental oxygen delivery; ERCP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ERCP patients monitored using currently marketed smart biteblock o2
  Interventions: Device: monitored using currently marketed smart biteblock o2
- 2 (Experimental): ERCP patients monitored using experimental biteblock delivering up to 10 lit/min oxygen
  Interventions: Device: monitored using investigational smart biteblock

INTERVENTIONS:
Device: monitored using currently marketed smart biteblock o2 — oral nasal CO2 monitoring and oxygen delivery
  Arms: 1
Device: monitored using investigational smart biteblock — monitored during ERCP procedure with nasal CO2 sampling and oral oxygen delivery at a flow rate up to 10 lit/min
  Arms: 2

SUMMARY:
The study hypothesis is that a modified smart bite block system can deliver up to 10 liters/minute of supplemental oxygen orally with the CO2 monitoring performance substantially equivalent to the currently marketed smart bite block that delivers oxygen up to 5 liters/minute

ELIGIBILITY:
Inclusion Criteria:

* For the Adults Bite Bloc:Adults >18 years old and able to understand and give consent per the Ethics committee requirements,or younger patients requiring an Adult size Bite Bloc in the opinion of the PI for whom the legal guardians consented for the participation of the trial.
* Patients consented or which their legal guardians consented for the participation of this trial.
* Clinical need to use a Bite Bloc to maintain an open mouth and protect the endoscope.
* Pediatric patients:patients with small mouth that the PI thinks require a Pediatric Bite Bloc (36 French),which their legal guardians consented for the participation of this trial.

Exclusion Criteria:

* Patients who are pregnant.
* Patients who in the opinion of the investigator should not participate.
* For Pediatric Bite Bloc:patients who need an Adult Bite Bloc to the investigators opinion or above the age of 12.
* Patients receiving oral or intravenous anticoagulants other than Aspirin or Plavix.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
EtCO2 measurement on the investigational device is equivalent to measurement on the control device | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: DAVID GOZAL, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel